CLINICAL TRIAL: NCT06131216
Title: Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-2022 Injection Alone or in Combination With Other Anti-tumor Treatments in Patients With Advanced Malignant Tumors
Brief Title: Phase I Study of SHR-2022 Injection in the Treatment of Patients With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2022-I-101
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Advanced Malignant Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-2022 Injection (Experimental)
  Interventions: Drug: SHR-2022 Injection

INTERVENTIONS:
Drug: SHR-2022 Injection — SHR-2022 Injection is administered by intravenous (IV) infusion

SUMMARY:
To evaluate the safety and tolerability of SHR-2022 in patients with advanced malignancies and to determine MTD or MAD versus RP2D

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this study, signed informed consent, compliance is good, can cooperate with follow-up
2. Age 18-80 years old (including both ends), both male and female
3. Subjects with advanced or metastatic malignant tumors confirmed by pathological tissue or cytology, and who have failed previous standard treatments, are intolerant to standard treatments, or have no standard treatments
4. Have measurable lesions
5. ECOG PS score: 0-1
6. Have a life expectancy of at least 3 months
7. The functional level of the major organs must meet the requirements
8. Fertile female patients must have a serum pregnancy test within 7 days before the first medication and the result is negative; And must be non-lactating

Exclusion Criteria:

1. Central nervous system metastasis or meningeal metastasis with clinical symptoms
2. Spinal cord compression that has not been treated radically by surgery and/or radiotherapy
3. Patients with uncontrolled tumor-related pain as judged by the investigator
4. A third space effusion with uncontrolled pleural effusion, pericardial effusion, or peritoneal effusion, as determined by the investigator
5. Systemic antitumor therapy was administered within 28 days prior to treatment in the first study
6. Surgical procedures requiring tracheal intubation and general anesthesia were performed within 28 days prior to the initial study, diagnostic or superficial surgery was performed within 7 days prior to the initial study, or elective surgery was expected during the trial period
7. Received within 28 days prior to the first investigational dose Non-radical chest radiation therapy of 30Gy received within 24 weeks prior to initial dosing. Patients receiving 30Gy of chest radiation therapy, and those receiving palliative radiation ≤30Gy within 14 days prior to the first dose
8. The AE caused by previous anti-tumor therapy did not recover to CTCAE v5.0 grade evaluation ≤1
9. Live attenuated vaccines were used within 28 days prior to administration in the first study or were expected to be required during the study treatment
10. Systemic immunosuppressive therapy was administered within 14 days prior to the first study
11. Accompanied by interstitial pneumonia or interstitial lung disease
12. Patients with a history of autoimmune disease
13. The first study studied patients with clinically significant bleeding symptoms or bleeding tendency within 3 months before medication
14. The first study was conducted in subjects with severe cardiovascular and cerebrovascular disease within 6 months prior to medication
15. Arterial/venous thrombosis events occurred within 3 months prior to initial administration
16. The first study studied any other malignancy within 5 years prior to medication
17. A known history of severe allergic reactions to the investigational drug and its principal formulation ingredients
18. Have a history of immune deficiency or organ transplantation, and have active hepatitis B or C
19. Severe infection within 4 weeks prior to the first dose
20. Patients with active pulmonary tuberculosis within 1 year prior to enrollment were found by history or CT examination
21. The presence of other serious physical or mental illness, known alcohol or drug dependence, abnormal laboratory tests, and other factors that may increase the risk of participating in the study or interfere with the study results; And any other conditions that the investigator deems inappropriate for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 3 years
Severity of adverse events | up to 3 years
MTD | up to 3 years
RP2D | up to 3 years

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | up to 3 year
Maximum concentration (Cmax) | up to 3 year
Receptor Occupancy（OR） of SHR-2022 | up to 3 year
Anti-drug antibody (ADA) of SHR-2022 | up to 3 year
Objective response rate (ORR) | up to 3 year

IPD SHARING:
Plan to Share IPD: Undecided